CLINICAL TRIAL: NCT03674307
Title: Canadian-Australasian Randomised Trial of Screening Kidney Transplant Candidates for Coronary Artery Disease
Brief Title: Screening for Asymptomatic Coronary Artery Disease in Kidney Transplant Candidates
Acronym: CARSK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Principal Investigator, John Gill, Professor of Medicine, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: H16-01335_CARSK
Record Dates: First submitted 2018-09-05; First posted 2018-09-17 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Diseases; End Stage Renal Disease; Kidney Transplantation; Dialysis Related Complication
MeSH Terms: conditions — Cardiovascular Diseases; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No screening (Experimental): No further screening for asymptomatic coronary artery disease after wait-list entry
  Interventions: Other: No screening
- Regular screening (Active Comparator): Regular (yearly or 2nd yearly) screening for asymptomatic coronary artery disease after wait-list entry
  Interventions: Other: Regular Screening

INTERVENTIONS:
Other: No screening — No further screening for asymptomatic coronary artery disease after wait-list entry
  Arms: No screening
Other: Regular Screening — Annual or second-yearly screening for asymptomatic coronary artery disease after wait-list entry
  Arms: Regular screening

SUMMARY:
The Canadian Australasian Randomized Trial of Screening Kidney Transplant Candidates for Coronary Artery Disease (CARSK) will test the hypothesis that eliminating the regular use of non-invasive screening tests for CAD AFTER waitlist activation is not inferior to regular (i.e., annual) screening for CAD during wait-listing for the prevention of Major Adverse Cardiac Events. Secondary analyses will assess the impact of screening on the rate of transplantation, and the relative cost-effectiveness of screening.

DETAILED DESCRIPTION:
Cardiovascular disease is the commonest cause of death while on the kidney transplant waiting list and after transplantation. Current standard care involves screening for coronary artery disease prior to waitlist entry, then every 1-2 years, according to perceived risk, until transplanted. The aim of screening is two-fold. Firstly to identify patients with asymptomatic coronary disease to enable either correction, by bypass surgery or angioplasty, or removal of the patient from the list, with the ultimate aim of preventing premature cardiovascular mortality at the time of, or soon after kidney transplantation. Secondly, from a societal perspective, to prevent mis-direction of scarce donor organs into recipients who experience early mortality. This current screening strategy is not evidence based, has substantial known and potential harms, and is very costly. Two major issues of uncertainty require addressing in sequence: (1) whether to periodically screen asymptomatic wait-listed patients for occult coronary artery disease; and (2) whether to revascularise coronary stenoses in asymptomatic patients prior to transplantation. The CARSK study seeks to address the first of these 2 issues.

CARSK aims to

1. Test the hypothesis that after screening for wait list entry, no further screening for coronary artery disease (CAD) is non-inferior to the current standard care which is screening all asymptomatic wait-listed patients for CAD at regular intervals.
2. Compare the benefits and costs of not screening versus regular CAD screening from a health system perspective.

ELIGIBILITY:
Inclusion Criteria:

1. adults aged 18 years of age or older
2. Dialysis-dependent kidney failure and currently being assessed for OR active on the kidney transplant waiting list
3. expected to require further screening for CAD prior to transplantation (by current standard of care);
4. able to give consent;
5. anticipated to undergo transplantation more than 12 months from date of enrolment

Exclusion Criteria:

1. patients with signs or symptoms suggestive of uncontrolled cardiac disease such as unstable coronary syndromes, decompensated heart failure, uncontrolled arrhythmia, and severe valvular heart disease;
2. patients who "on-hold" for transplantation due to a medical problem;
3. patients with other solid organ transplants;
4. multi-organ transplant candidates (e.g. kidney-pancreas transplant candidates);
5. patients with planned living donor transplant;
6. patients unable to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3306 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
MACE | The investigators will analyse time to first MACE event for the duration of the trial (60 months), depending on patient's date of transplant. Follow-up will be 12 months posttransplant. Maximum follow-up is 72 months.
  Primary efficacy: major adverse cardiac event (MACE), defined as any of the following: cardiovascular death, myocardial infarction, emergency revascularisation, hospitalisation with unstable angina.
  The outcome will be assessed by:
  1. Notification to the transplant coordinators when patients are admitted in hospital (this is the usual standard of care in waitlisted patients).
  2. The trial coordinator will gather electronic medical records, letters, procedure notes, and will fill in the relevant case record form on the REDCap database (managed by Sydney local health district). All data are encrypted and stored on servers at SLHD, where it is backed up.
  3. Patients will be followed up 6-monthly (alternating by phone and clinic visits) where trial coordinators will discuss any hospitalisation with the patients.

SECONDARY OUTCOMES:
All-cause death | Between 24 and 72 months, depending on patient's date of transplant. Follow-up will be 12 months posttransplant
  Death due to any cause
Emergency revascularisation | Between 24 and 72 months, depending on patient's date of transplant. Follow-up will be 12 months posttransplant
  Urgent, symptom-driven revascularisation for coronary artery disease
Stroke | Between 24 and 72 months, depending on patient's date of transplant. Follow-up will be 12 months posttransplant
  Stroke
Health related quality of life | Between 24 and 72 months, depending on patient's date of transplant. Follow-up will be 12 months posttransplant
  health related quality of life as measured by EQ5D and/or KDQOL 36
Time of wait-listing | Between 24 and 72 months, depending on patient's date of transplant. Follow-up will be 12 months posttransplant
  Time off the wait-list
Cost effectiveness | The analysis will take place at the end of the study. This outcome will be followed up for 5 years.
  Economic evaluation of the cost effectiveness of the trial from a health system perspective.
  Data on resource use will be obtained in two ways. First through identification of tests, procedures and doctor's visits related to cardiac and renal management for all study participants from randomisation to study end as recorded in the patient diaries and trial case report forms. Second, Australian participants will have their records linked to the Admitted Patient Data Collection, Emergency Department Data Collection, and through Medicare for all Medicare Benefits Schedule (MBS) outpatient visits, procedures and the Pharmaceutical Benefits Scheme (PBS) for medicines.
Incidence of transplantation | Between 24 and 72 months, depending on patient's date of transplant. Follow-up will be 12 months posttransplant
  incidence of transplantation between the two arms
Incidence of permanent removal from wait list for cardiac causes | Between 24 and 72 months, depending on patient's date of transplant. Follow-up will be 12 months posttransplant
  incidence of permanent removal from the wait list due to cardiac causes between the two arms
Cancellation of transplantation due to coronary artery disease | Between 24 and 72 months, depending on patient's date of transplant. Follow-up will be 12 months posttransplant
  incidence of cancellation of transplantation due to coronary artery disease
Cardiovascular death | Between 24 and 72 months, depending on patient's date of transplant. Follow-up will be 12 months posttransplant
  incidence of cardiovascular death

CONTACTS AND LOCATIONS:
Overall Officials: Jagbir Gill, MD, Principal Investigator — University of British Columbia
Locations (22):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - The George Washington University, Washington D.C., District of Columbia
- Canada (14):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Dalhousie University, Halifax, Nova Scotia
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Kingston Health Science Centre, Kingston, Ontario
  - London Health Science Centre, London, Ontario
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - CHU de Quebec-Universite Laval's L'Hotel-Dieu de Quebec, Laval, Quebec
  - University of Montreal, Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Universite de Montreal, Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - St. Paul's Hospital, University of Saskatchewan, Saskatoon, Saskatchewan
- Charité Universitätsmedizin, Berlin, Germany
- United Kingdom (5):
  - Sussex Brighton R&D, Brighton
  - King's College Hospital NHS Foundation Trust, Brixton
  - Epsom and St Helier University Hospitals NHS Trust, Carshalton
  - Barts Health NHS Trust, London
  - St George's University Hospital NHS Trust Foundation, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ying T, Gill J, Webster A, Kim SJ, Morton R, Klarenbach SW, Kelly P, Ramsay T, Knoll GA, Pilmore H, Hughes G, Herzog CA, Chadban S, Gill JS. Canadian-Australasian Randomised trial of screening kidney transplant candidates for coronary artery disease-A trial protocol for the CARSK study. Am Heart J. 2019 Aug;214:175-183. doi: 10.1016/j.ahj.2019.05.008. Epub 2019 May 22. PMID 31228771

DOCUMENTS (1):
  • Study Protocol (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT03674307/Prot_000.pdf